CLINICAL TRIAL: NCT02148874
Title: Immune Responses to the Flu Shot During Pregnancy
Status: Completed | Type: Observational
Sponsor: Lisa Christian (Other)
Responsible Party: Sponsor-Investigator, Lisa Christian, Assistant Professor, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2008H0260
Record Dates: First submitted 2014-05-23; First posted 2014-05-28 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Pregnancy
Keywords: pregnant; flu shot; influenza; vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum whole blood plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Flu Shot: pregnant women receive a seasonal influenza virus vaccination
  Interventions: Biological: influenza virus vaccination

INTERVENTIONS:
Biological: influenza virus vaccination — comparison of immune responses to the flu vaccine in obese and non-obese populations
  Other Names: flu shot; influenza shot; flu vaccine

SUMMARY:
This study will examine effects of everyday life stress and obesity on immune responses to influenza virus vaccine (the flu shot) during pregnancy. Following vaccination, antibody levels against influenza (the flu) increase. Higher antibody levels indicate better immune protection from influenza. In addition to providing protection from the flu for yourself, being vaccinated during pregnancy may protect your baby from the flu during the first six months of life during which time infants cannot be vaccinated. Our primary goals are to determine whether greater life stress and obesity reduce 1) antibody responses to the flu shot in women and 2) antibody levels in the newborn at the time of delivery.

ELIGIBILITY:
Inclusion Criteria:

* less than 29 weeks pregnant
* ages 18-42
* planning to deliver at The Ohio State University Wexner Medical Center

Exclusion Criteria:

* prior serious adverse reaction to seasonal influenza vaccine

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: community sample, prenatal clinic
Sampling Method: Non-Probability Sample
Enrollment: 287 (Actual)
Dates: Start 2013-10; Primary Completion 2017-05 (Actual); Study Completion 2019-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M. Christian, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Derived] Christian LM, Beverly C, Mitchell AM, Karlsson E, Porter K, Schultz-Cherry S, Ramilo O. Effects of prior influenza virus vaccination on maternal antibody responses: Implications for achieving protection in the newborns. Vaccine. 2017 Sep 18;35(39):5283-5290. doi: 10.1016/j.vaccine.2017.05.050. Epub 2017 Aug 1. PMID 28778612
- See also: For more information or to apply — http://stressandpregnancy.osumc.edu/Pages/default.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We enrolled 287 pregnant women between October 2013 and March 2017 at The Ohio State University Wexner Medical Center. Participants were recruited through prenatal clinics at Ohio State, campus newsletters and advertisements, and community online advertisements.
Groups:
- Non-Obese: Pregnant women with a pre-pregnancy BMI 18.5-29.9.
- Obese: Pregnant women with a pre-pregnancy BMI 30.0-50.0
Period: Overall Study
Arm/Group | Non-Obese | Obese
Started | 201 | 86
Completed | 194 | 84
Not Completed | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-Obese | Obese | Total
Number analyzed (Participants) | 201 | 86 | 287
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 201 | 86 | 287
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 201 | 86 | 287
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 10
  Not Hispanic or Latino | 195 | 82 | 277
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 38 | 33 | 71
  White | 150 | 49 | 199
  More than one race | 8 | 3 | 11
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 201 | 86 | 287

OUTCOME MEASURES:

1. Primary Outcome: Maternal HAI Antibody Titers
Description: Maternal influenza antibody titers from hemagglutination inhibition (HAI) assay
Time Frame: 30-days after influenza vaccination
Population: Pregnant women with antibody titer data at 30 days post vaccination. Analyses include all women with available antibody titer data at the necessary time points.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Non-Obese | Obese
Number analyzed (Participants) | 188 | 75
Titer
  A/H1N1 Strain | 55.9 [43.0 to 72.5] | 59.8 [41.1 to 87.0]
  A/H3N2 Strain | 78.5 [60.9 to 101.1] | 74.0 [48.9 to 112.1]
  B/Massachusetts Strain | 17.3 [13.9 to 21.6] | 22.3 [15.2 to 32.8]
  B/Brisbane Strain | 17.8 [14.4 to 22.1] | 20.8 [14.1 to 30.6]
Statistical Analysis 1: Comparison: Non-Obese vs Obese; Statistical analysis for influenza strain A/H1N1; Test type: Superiority; p = 0.84, Regression, Logistic; Cumulative logistic regression model; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.64 to 1.73] — Cumulative logistic regression model, OR for obese vs. non-obese. Model adjusted for mother's age, parity, gestational age at vaccination, vaccination season, and prior year vaccination (Y/N)
Statistical Analysis 2: Comparison: Non-Obese vs Obese; Statistical analysis for influenza strain A/H3N2; Test type: Superiority; p = 0.79, Regression, Logistic; Cumulative logistic regression model; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.65 to 1.75] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Non-Obese vs Obese; Statistical analysis for influenza strain B/Massachusetts; Test type: Superiority; p = 0.43, Regression, Logistic; Cumulative logistic regression model; Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.71 to 2.24] — Cumulative logistic regression model, OR for obese vs. non-obese. Model adjusted for mother's age, parity, gestational age at vaccination, vaccination season, and prior year vaccination (Y/ N)
Statistical Analysis 4: Comparison: Non-Obese vs Obese; Statistical analysis for influenza strain B/Brisbane; Test type: Superiority; p = 0.77, Regression, Logistic; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.63 to 1.87] — [estimate comment as in outcome 1, analysis 3]

2. Primary Outcome: Maternal HAI Antibody Titers
Description: Maternal influenza antibody titers from hemagglutination inhibition (HAI) assay
Time Frame: at delivery
Population: Pregnant women with antibody titer data at delivery. Analyses include all women with available antibody titer data at the necessary time points.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Non-Obese | Obese
Number analyzed (Participants) | 181 | 79
Titer
  A/H1N1 Strain | 23.5 [18.5 to 29.8] | 32.5 [22.6 to 46.8]
  A/H3N2 Strain | 31.6 [24.8 to 40.4] | 32.7 [22.3 to 47.8]
  B/Massachusetts Strain | 10.3 [8.6 to 12.3] | 16.3 [11.9 to 22.2]
  B/Brisbane Strain | 8.4 [7.2 to 9.9] | 11.4 [8.5 to 15.4]
Statistical Analysis 1: Comparison: Non-Obese vs Obese; Statistical analysis for influenza strain A/H1N1; Test type: Superiority; p = 0.20, Regression, Logistic; Cumulative logistic regression model; Odds Ratio (OR) = 1.39, 95% CI 2-sided [0.84 to 2.32] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Non-Obese vs Obese; Statistical analysis for influenza strain A/H3N2; Test type: Superiority; p = 0.74, Regression, Logistic; Cumulative logistic regression model; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.66 to 1.80] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Non-Obese vs Obese; Statistical analysis for influenza strain B/Massachusetts; Test type: Superiority; p = 0.04, Regression, Logistic; Cumulative logistic regression model; Odds Ratio (OR) = 1.89, 95% CI 2-sided [1.04 to 3.44] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Non-Obese vs Obese; Statistical analysis for influenza strain B/Brisbane; Test type: Superiority; p = 0.13, Regression, Logistic; Cumulative logistic regression model; Odds Ratio (OR) = 1.63, 95% CI 2-sided [0.87 to 3.04] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Infant HAI Antibody Titers
Description: Infant influenza antibody titers from hemagglutination inhibition (HAI) assay
Time Frame: cord blood at delivery
Population: Cord blood from participating pregnant women with cord blood data available. There was only one cord blood sample per participant in this study.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Non-Obese | Obese
Number analyzed (Participants) | 165 | 69
Titer
  A/H1N1 Strain | 95.4 [78.6 to 115.7] | 78.4 [54.7 to 112.4]
  A/H3N2 Strain | 155.5 [125.2 to 192.9] | 118.2 [80.8 to 172.8]
  B/Massachusetts Strain | 139.0 [113.0 to 170.9] | 157.0 [114.1 to 215.9]
  B/Brisbane Strain | 128.8 [106.2 to 156.3] | 99.1 [68.5 to 143.3]
Statistical Analysis 1: Comparison: Non-Obese vs Obese; Statistical analysis for influenza strain A/H1N1; Test type: Superiority; p = 0.64, Regression, Logistic; Cumulative logistic regression model; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.53 to 1.48] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Non-Obese vs Obese; Statistical analysis for influenza strain A/H3N2; Test type: Superiority; p = 0.67, Regression, Logistic; Cumulative logistic regression model; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.53 to 1.50] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Non-Obese vs Obese; Statistical analysis for influenza strain B/Massachusetts; Test type: Superiority; p = 0.14, Regression, Logistic; Cumulative logistic regression model; Odds Ratio (OR) = 1.47, 95% CI 2-sided [0.88 to 2.46] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Non-Obese vs Obese; Statistical analysis for influenza strain B/Brisbane; Test type: Superiority; p = 0.25, Regression, Logistic; Cumulative logistic regression model; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.44 to 1.24] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from enrollment up until delivery of the infant. This time frame varied from 3-8 months depending on gestational age at enrollment.
Arm/Group | Non-Obese | Obese
All-Cause Mortality (participants affected / at risk) | 0/201 | 0/86
Serious Adverse Events (participants affected / at risk) | 0/201 | 0/86
Other Adverse Events (participants affected / at risk) | 0/201 | 0/86

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-19): https://cdn.clinicaltrials.gov/large-docs/74/NCT02148874/Prot_SAP_000.pdf